CLINICAL TRIAL: NCT04987177
Title: Relationship Among Manual Wheelchair Workload, Speed, Energy Expenditure, and Propulsion Mechanics
Brief Title: Effect of Manual Wheelchair Propulsion Workload on Speed, Energy Expenditure, and Propulsion Mechanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachel Cowan, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300007513
Record Dates: First submitted 2021-07-16; First posted 2021-08-03 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Healthy Participants
Keywords: workload; wheelchair; biomechanics; energy expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Workload conditions to be tested (Experimental): The intervention is the external workload a participant propels against. Participants will propel against N=20 different external workloads.External workload will be controlled by the wheelchair ergometer.
  Interventions: Other: Workload of Manual Wheelchair Propulsion

INTERVENTIONS:
Other: Workload of Manual Wheelchair Propulsion — Participants will complete 20 one-minute manual wheelchair propulsion bouts. Each one minute propulsion bout will be followed by a 2 minute rest period. Each propulsion bout will be at a different workload. After every 10 propulsion bouts, participants will be provided with an extended rest period (5 to 30 minutes). For each participant, the maximum workload to be tested is based on their estimated maximum workload. Estimate maximum workload is based on the HR-Workload relationship documented during a prior sub maximal test to 80% of age adjusted maximum heart rate.

SUMMARY:
The first purpose of this study is to characterize the relationship among propulsion workload, self-selected propulsion speed, and propulsion kinetics/kinematics.

The second purpose is to assess the between days repeatability/reliability of the above outcomes.

There are no hypothesis

This is a repeated measures clinical trial. All participants will complete the following: 1) Acclimation to propelling a manual wheelchair on a wheelchair ergometer; 2) Graded exercise test on the wheelchair ergometer to 80% of age adjusted estimated maximal heart rate; and 3) N=20 one minute propulsion bouts on the wheelchair ergometer.

DETAILED DESCRIPTION:
Participants will complete two visits in a 14 day period. Visit 1 will require 3-4 hours. Visit 2 will require 2-3 hours.

During visit 1 participant will complete: 1) Acclimation to propelling a manual wheelchair on a wheelchair ergometer; 2) Graded exercise test on the wheelchair ergometer to 80% of age adjusted estimated maximal heart rate; and 3) N=20 one minute propulsion bouts on the wheelchair ergometer.

During visit 2 participants will repeat the N=20 one minute propulsion bouts on the wheelchair ergometer.

Wheelchair ergometer propulsion acclimation: Participants will complete a minimum of 2 minutes of wheelchair propulsion to acclimate. Additional propulsion time will be completed as needed. Propulsion workload will be varied during the acclimation. Acclimation propulsion may be repeated as needed during study participation.

Submaximal wheelchair ergometer test protocol: Participants will rest quietly in the wheelchair for several minutes. After resting, participants will begin propelling at a comfortable speed at a low initial workload. Workload will be increased every minute. Propulsion speed will remain constant across all workloads. Test will end when participants reach 80% of age adjusted estimated maximum heart rate.

Wheelchair propulsion workload assessment: Participants will complete 20 one-minute propulsion bouts at a self-selected speed. Each one minute propulsion bout will be followed by a 2 minute rest period. Each propulsion bout will be at a different workload. After the first 10 propulsion bouts, participants will be provided with an extended rest period (5 to 30 minutes). For each participant, the maximum workload to be tested is based on their estimated maximum workload. Estimate maximum workload is based on the Heart Rate-Workload relationship documented during the submaximal test.

The workloads of the N=20 propulsion bouts will be divided into two groups of N=10 (Group A and Group B). The total workload of each group will be equal. Within each group, workload sequence is fixed and arranged in a non-ascending or descending order. Completion order of the groups will be counterbalanced within sex. Within participants, completion order will be counterbalanced across days

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* cleared to participate in physical activity as determined by the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
* self-reported ability to propel a manual wheelchair
* not currently disabled

Exclusion Criteria:

* no additional exclusion criteria if otherwise eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Self-Selected Speed (meters per second) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average linear propulsion speed during each completed propulsion cycle (i.e. contact+recovery) averaged across all completed propulsion cycles in the specified time frame.
Average Rolling Resistance (Newtons) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average rolling resistance during each completed propulsion cycle (i.e. contact+recovery) averaged across all completed propulsion cycles in the specified time frame.

SECONDARY OUTCOMES:
Number of completed propulsion cycles used to generate the outcomes of interest | Seconds 20 to 40 of each 1 minute propulsion bout
  The number of complete propulsion cycles occurring in the specified time frame. A complete propulsion cycle is defined as beginning with the onset of contact with the pushrim and ending with the onset of contact of the next propulsion cycle. A propulsion cycle includes contact and recovery.
Average resultant force (Newtons) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average resultant force during the contact phase of each completed propulsion cycle averaged across all completed propulsion cycles in the specified time frame.
Average rate of rise of resultant force (Newtons per second squared) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average rate of rise of resultant force during the contact phase of each completed propulsion cycle averaged across all completed propulsion cycles in the specified time frame.
Average push frequency (pushes per minute) | Seconds 20 to 40 of each 1 minute propulsion bout
  For the specified time frame, the total number of completed propulsion cycles divided by the time to complete all the propulsion cycles in seconds multiplied by 60 seconds.
Average push length (Degrees) | Seconds 20 to 40 of each 1 minute propulsion bout
  The distance over which a propulsive torque is applied to the pushrim during the contact phase of each complete propulsion cycle averaged across all completed propulsion cycles in the specified time frame.
Average propulsive torque (Newton meter) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average propulsive torque during the contact phase of each completed propulsion cycle averaged across all completed propulsion cycles in the specified time frame.
Average push power output (Watts) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average power during the contact phase of each each completed propulsion cycle averaged across all completed propulsion cycles in the time frame of interest. Push power output represents the energy the person applies to the pushrim during the contact phase.
Average total work per push (Joules) | Seconds 20 to 40 of each 1 minute propulsion bout
  Total work during the contact phase of each completed propulsion cycle averaged across all completed propulsion cycles in the time frame of interest.
Average external power output (Watts) | Seconds 20 to 40 of each 1 minute propulsion bout
  Average external power output during the entire propulsion cycle (i.e. contact and recovery) averaged across all completed propulsion cycles in the specified time frame. External power output represents the energy expended by the user-wheelchair system.
Frequency of each unique propulsion pattern | Seconds 20 to 40 of each 1 minute propulsion bout
  For each complete propulsion cycle during the specified time frame, the recovery pattern will be classified into one of 5 categories: semi-circular, arcing, single loop, double loop, or indeterminate. The number of cycles and overall percentage in each category will be reported. Overall percentage is defined as [number of cycles in a category/total number of cycles * 100].

CONTACTS AND LOCATIONS:
Locations (1):
- UAB/Lakeshore Research Colaborative Building, Homewood, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soleymani H, Cowan R. Relationship between rolling resistance, preferred speed, and manual wheelchair propulsion mechanics in non-disabled adults. Disabil Rehabil Assist Technol. 2024 Jul;19(5):1980-1991. doi: 10.1080/17483107.2023.2239297. Epub 2023 Jul 26. PMID 37493253